CLINICAL TRIAL: NCT04965532
Title: Second Affiliated Hospital Zhejiang University School of Medicine
Brief Title: Residual Neuromuscular Block of Rocuronium in Chemotherapy Patients Under Sevoflurane Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-046
Record Dates: First submitted 2021-07-06; First posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-06

CONDITIONS: Chemotherapeutic Toxicity
MeSH Terms: interventions — Anesthesia, Inhalation; Propofol; Anesthesia, Intravenous

STUDY DESIGN:
Intervention Model Description: Eighty patients undergoing liver radiofrequency ablation surgery under elective general anesthesia were selected, of whom 40 received preoperative adjuvant chemotherapy and the other 40 were nonchemotherapy patients, who were divided by randomization according to the method of anesthesia maintenance, respectively.Chemotherapy patients were divided into PC group with 20 cases using all intravenous anesthesia and SC group with 20 cases using sevoflurane anesthesia.The nonchemotherapy patients were divided into PN group with 20 cases using all intravenous anesthesia and Sn group with 20 cases using sevoflurane anesthesia.
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- chemotherapy patients using sevoflurane anesthesia (Experimental): Following induction of anesthesia and laryngeal mask placement, anesthesia will be maintained by inhalation of sevoflurane (approximately 1.3 × minimum alveolar concentration) and IV fentanyl according to clinical need.
  Interventions: Drug: sevoflurane anesthesia
- chemotherapy patients using total intravenous anesthesia (Active Comparator): Following induction of anesthesia and laryngeal mask placement, maintenance of anesthesia will consist of target-controlled infusion of propofol at a plasma target concentration of 1.5-3.0µg/ml and IV fentanyl according to clinical need.
  Interventions: Drug: Propofol Injection
- nonchemotherapy patients using sevoflurane anesthesia (Active Comparator): Following induction of anesthesia and laryngeal mask placement, anesthesia will be maintained by inhalation of sevoflurane (approximately 1.3 × minimum alveolar concentration) and IV fentanyl according to clinical need.
  Interventions: Drug: sevoflurane anesthesia
- nonchemotherapy patient using total intravenous anesthesia (Active Comparator): Following induction of anesthesia and laryngeal mask placement, maintenance of anesthesia will consist of target-controlled infusion of propofol at a plasma target concentration of 1.5-3.0µg/ml and IV fentanyl according to clinical need.
  Interventions: Drug: Propofol Injection

INTERVENTIONS:
Drug: sevoflurane anesthesia — Sevoflurane enhances the effects of rocuronium and significantly prolongs the duration of action of rocuronium and the time to recovery.
  Other Names: inhalation anesthesia
  Arms: chemotherapy patients using sevoflurane anesthesia; nonchemotherapy patients using sevoflurane anesthesia
Drug: Propofol Injection — Propofol is most commonly used for intravenous anesthesia. In contrast to sevoflurane, propofol has no effects on rocuronium.
  Other Names: intravenous anesthesia
  Arms: chemotherapy patients using total intravenous anesthesia; nonchemotherapy patient using total intravenous anesthesia

SUMMARY:
Chemotherapy causes motor nerve dysfunction and degeneration that may alter the response to neuromuscular blocking drugs. To analyse the risk of residual neuromuscular block (RNMB) induced by rocuronium given in standard doses to patients who undergo chemotherapy within three months.

DETAILED DESCRIPTION:
Rocuronium, as a non depolarizing muscle relaxant with medium time effect, takes effect rapidly. It is an ideal neuromuscular blocker to replace succinylcholine for induction of tracheal intubation and maintenance of muscle relaxant under general anesthesia. Sevoflurane is widely used in clinic because of its low blood gas partition coefficient, rapid and stable induction and recovery, easy adjustment of anesthesia depth and strong controllability. In addition, the number of patients receiving preoperative adjuvant chemotherapy for malignant tumors is increasing year by year in China. The commonly used chemotherapy drugs, such as paclitaxel, platinum, vinorelbine, etc., have dose-dependent peripheral neurotoxicity. Therefore, to explore and study the influence of pathophysiological changes of patients receiving chemotherapy on the neuromuscular relaxation effect of sevoflurane combined with non depolarizing neuromuscular blockers, It is very important for anesthesia, resuscitation and perioperative management of chemotherapy patients. The purpose of this study is to reveal the effect of sevoflurane on rocuronium neuromuscular blockade in chemotherapy patients by comparing the difference of rocuronium neuromuscular blockade effect of sevoflurane and total intravenous anesthesia in chemotherapy patients and non chemotherapy patients, and to provide information for more safe and rational application of rocuronium in clinical anesthesia of chemotherapy patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients classified as American Society of Anesthesiology physical status (ASA PS) classes I, II or III
* Aged between 18 and 70 years
* Scheduled for radiofrequency ablation of liver tumours under general anaesthesia with an expected surgery duration shorter than 60min

Exclusion Criteria:

* Allergy to rocuronium
* Myasthenia gravis
* Guillain-Barre ́ syndrome
* Duchenne muscular dystrophy or similar
* Receiving drugs that might interfere with the neuromuscular transmission or the response to neuromuscular blockers, such as some anticonvulsants and antibiotics

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Muscle relaxation recovery index | The first 90 min following intravenous injection of rocuronium
  Time interval from 25% recovery to 75% recovery of the first twitch in the TOF stimulation pattern

SECONDARY OUTCOMES:
Onset time of muscle relaxation | The first 90 min following intravenous injection of rocuronium
  Time interval from the completion of intravenous injection of rocuronium to the maximal depression of the first twitch in the TOF stimulation pattern

OTHER OUTCOMES:
Clinical duration of muscle relaxation | The first 90min following intravenous injection of rocuronium
  Time interval from the completion of intravenous injection of rocuronium to 25% recovery of the first twitch in the TOF stimulation pattern
TOF ratio | 10min following intravenous injection of rocuronium
  Dividing the amplitude of the fourth response by the amplitude of the first response
T1 amplitude | 10min following intravenous injection of rocuronium
  The amplitude of the first twitch to TOF stimulation
TOF ratio | 20min following intravenous injection of rocuronium
  Dividing the amplitude of the fourth response by the amplitude of the first response
T1 amplitude | 20min following intravenous injection of rocuronium
  The amplitude of the first twitch to TOF stimulation
TOF ratio | 30min following intravenous injection of rocuronium
  Dividing the amplitude of the fourth response by the amplitude of the first response
T1 amplitude | 30min following intravenous injection of rocuronium
  The amplitude of the first twitch to TOF stimulation
TOF ratio | 40min following intravenous injection of rocuronium
  Dividing the amplitude of the fourth response by the amplitude of the first response
T1 amplitude | 40min following intravenous injection of rocuronium
  The amplitude of the first twitch to TOF stimulation
TOF ratio | 50min following intravenous injection of rocuronium
  Dividing the amplitude of the fourth response by the amplitude of the first response
T1 amplitude | 50min following intravenous injection of rocuronium
  The amplitude of the first twitch to TOF stimulation
TOF ratio | 60min following intravenous injection of rocuronium
  Dividing the amplitude of the fourth response by the amplitude of the first response
T1 amplitude | 60min following intravenous injection of rocuronium
  The amplitude of the first twitch to TOF stimulation
TOF ratio | 70min following intravenous injection of rocuronium
  Dividing the amplitude of the fourth response by the amplitude of the first response
T1 amplitude | 70min following intravenous injection of rocuronium
  The amplitude of the first twitch to TOF stimulation
TOF ratio | 80min following intravenous injection of rocuronium
  Dividing the amplitude of the fourth response by the amplitude of the first response
T1 amplitude | 80min following intravenous injection of rocuronium
  The amplitude of the first twitch to TOF stimulation
TOF ratio | 90min following intravenous injection of rocuronium
  Dividing the amplitude of the fourth response by the amplitude of the first response
T1 amplitude | 90min following intravenous injection of rocuronium
  The amplitude of the first twitch to TOF stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Lili Fang, Dr., Principal Investigator — Second Affiliated Hospital Zhejiang University School of Medicine
Locations (2):
- China (2):
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - Quzhou People's Hospital, Quzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No